

**Procedure Title: TREAT GRX Study** 

Protocol

Doc Number: 104-09062

Revision: A 

## TREAT GRX STUDY SUMMARY

TITLE An Evaluation of Performance of the CorPath® GRX System in

Robotic-PCI during Acute STEMI

SHORT TITLE TREAT GRX Study

**DEVICE** CorPath® GRX System:

Bedside Unit consists of the Extended Reach Arm,

Robotic Drive, and single-use Cassette.

Interventional cockpit

Control console

**REGULATORY STATUS** The CorPath GRX System was granted 510(k) clearance

(K160121) on October 27, 2016.

**INDICATION FOR USE** The CorPath GRX System is intended for use in the remote

delivery and manipulation of guidewires and rapid exchange catheters, and remote manipulation of guide catheters during

percutaneous coronary and vascular procedures.

STUDY OBJECTIVE This study will evaluate the performance of the CorPath GRX

System in Robotic Primary PCI (RPPCI) in the treatment of

STEMI.

STUDY DESIGN This is a prospective, post-market, single-arm, multi-center,

observational study to evaluate the performance of the CorPath

GRX System during robotic-PCI for acute ST elevation

myocardial infarction (STEMI).

PRINCIPAL INVESTIGATOR Salvatore F. Mannino, DO, MA, FACC, FSCAI

Interventional Director, Short Term Mechanical Circulatory

Support Program

WellStar Health System

55 Whitcher St Suite 350

Marietta, GA 30060 USA

**SAMPLE SIZE** Up to 100 subjects shall be enrolled in the study.

**INVESTIGATIONAL SITES** A maximum of five (5) sites may participate.



**Procedure Title: TREAT GRX Study** 

Protocol

Doc Number: 104-09062

Revision: A 

**EVALUATION PERIOD** Estimated date of first patient enrolled: August 2020

Anticipated enrollment period: 12 months

Estimated date of last patient enrolled: August 2021

STUDY DURATION/ FOLLOW-UP PERIOD All subjects will be followed post-CorPath GRX PCI procedure

through 72-hours post-procedure or hospital discharge,

whichever occurs first.

SUBJECT POPULATION Subjects with a clinical indication of STEMI.

INCLUSION CRITERIA Candidates will be included in the study only if all the following

conditions are met:

• Age ≥18 and ≤ 80 years

Patients with STEMI<12 h of symptom onset</li>

Patient deemed appropriate for robotic-assisted PCI

 The subject has been informed of the nature of the study, agrees to its provisions, and has provided written

consent

EXCLUSION CRITERIA

Candidates will be excluded from the study if any of the following conditions are present:

- Cardiogenic shock
- Cardiac arrest
- Need for manual or mechanical thrombectomy
- Failure/inability/unwillingness to provide informed consent
- The Investigator determines that the subject or the coronary anatomy is not suitable for robotic-assisted primary PCI treatment

PRIMARY ENDPOINT

Time from Catheterization Lab Arrival to Device Activation (CLADA) by CorPath GRX System.



| Procedure Title: TREAT GRX Study Protocol | |
|-------------------------------------------|-----------------------|
| Doc Number: 104-09062 | |
| Revision: A | <b>Page</b> : 8 of 34 |

#### **SECONDARY ENDPOINTS**

## Freedom from MACE events

Completion of the STEMI procedure without in-hospital major adverse cardiovascular event MACE). MACE is defined as cardiac death, clinically driven target vessel revascularization (TVR) by repeat PCI, surgical bypass for any segment of the target vessel or stent thrombosis.

# First Medical Contact (FMC) to device activation time

Time at which the patient was first evaluated by Emergency Medical System (EMS) or Emergency Department arrival to device activation.

## Access to device activation

Time from initial sheath insertion to device activation.

#### Access to wire time

Defined as time measured from sheath insertion to crossing the lesion with the coronary guidewire.

# Overall procedure time

Defined as the time measured from sheath insertion to removal of the last device used to treat the culprit lesion.

# Fluoroscopy time

Total fluoroscopy time (min.) utilized during the procedure as recorded by the Imaging System.

## Patient radiation exposure

DAP (dose-area-product) and AK (air kerma) as recorded during the procedure.

#### Contrast fluid volume

Total contrast volume (mL/cc) used during the procedure.

## **Conversion to manual (Binary)**

Conversion from robotic technique to manual technique due to inability to successfully wire lesion or deliver first device.

## **Technical success**

Completion of the PCI procedure entirely robotically or with partial manual assistance.



**Procedure Title: TREAT GRX Study** 

Protocol

Doc Number: 104-09062

Revision: A 

Serious adverse events

All Serious Adverse Events (SAEs) from the start of the CorPath GRX procedure until the end of the study will be

summarized.

STUDY SPONSOR Corindus, Inc.

309 Waverley Oaks Road, Suite 105

Waltham, MA 02452 USA

MANUFACTURER Corindus, Inc.

309 Waverley Oaks Road, Suite 105

Waltham, MA 02452 USA

**DATA COORDINATING** 

CENTER

MedNet Solutions, Inc.

110 Cheshire Lane, Suite 300

Minnetonka, MN 55305

MONITORING SERVICE Corindus, Inc.

309 Waverley Oaks Road, Suite 105

Waltham, MA 02452 USA

STATISTICAL ANALYSIS

**SERVICES** 

**TBD**